CLINICAL TRIAL: NCT03205072
Title: Per-Oral Cholangioscopy in Liver Transplantation Patients
Brief Title: POCS in Liver Transplantation Patients
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: E7114
Record Dates: First submitted 2017-06-26; First posted 2017-07-02 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Liver Transplant; Complications
Keywords: ERCP; Per-Oral Cholangioscopy; Liver Transplantation; Spy Glass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Biopsies if needed at the discretion of the PI.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- ERCP & Spy Glass DS: Patients with cadaveric donor or live donor liver transplantation referred for ERCP in the setting of a clinical suspicion of post liver transplant bile duct strictures.
  Interventions: Device: Spy Glass DS

INTERVENTIONS:
Device: Spy Glass DS — The SpyScope™ DS Access and Delivery Catheter (SpyScope™ DS Catheter) is a sterile, single-use endoscope that enables access and delivery of accessories to targeted pancreaticobiliary anatomy and displays live video when connected to a Spy Glass DS Digital Controller.

SUMMARY:
A prospective, multi-center, non-randomized, observational, consecutive case series, which will compare Endoscopic Retrograde Cholangiopancreatoscopy (ERCP) and cholangioscopy with Spy Glass Digital System (DS) procedure at 5-10 centers.

DETAILED DESCRIPTION:
The objective of this study is to demonstrate the clinical utility of cholangioscopy with Spy Glass Digital System (DS) in cadaveric donor or live donor liver transplantation patients who are referred for ERCP in the setting of a clinical suspicion of post liver transplant bile duct stricture(s). A secondary study objective is to generate a hypothesis for a randomized controlled trial comparing ERCP alone to ERCP with Per- Oral Cholangioscopy (POCS) in patients referred for ERCP post liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Liver transplantation at least 1 month prior to POCS procedure
2. Abnormal Liver Function Tests (LFTs) and/or biliary obstructive symptoms
3. Prior cross sectional imaging (MRI and/or US and/or CT)
4. Suspicion of anastomotic biliary stricture(s)
5. Diameter of bile ducts deemed sufficient to accommodate cholangioscopy system based on baseline imaging
6. Willing and able to provide a written informed consent to participate in the study
7. Willing and able to comply with study procedures and follow-up schedule

Exclusion Criteria:

1. Contraindication for an ERCP per local standard of practice
2. Deemed contraindicated for POCS per local standard of practice
3. Prior biliary treatment of biliary anastomotic stricture
4. < 18 years old
5. Documented life expectancy of less than 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cadaveric donor or live donor liver transplantation patients referred for ERCP in the setting of a clinical suspicion of post-liver transplant bile duct stricture(s).
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-24 (Actual)

PRIMARY OUTCOMES:
Impact of Per-Oral Cholangioscopy on Patient Management | 12 Months
  To evaluate the impact of the addition of POCS to same setting ERCP on the recommended management of post-liver transplantation biliary complications.

SECONDARY OUTCOMES:
Technical Success | 12 Months
  Ability to visualize the duct/lesion of interest and, if applicable, ability to obtain POCS-guided biopsy adequate for histopathology.
Serious Adverse Events | 12 Months
  Serious Adverse Events (SAEs) including severity, onset, time to resolution, required interventions, relatedness to endoscopic devices and/or procedures and hospitalizations.
Number of biliary re-interventions | 12 Months
  Re-interventions may include but are not limited to repeat ERCP, repeat POCS, ultrasonography, stent exchanges, balloon dilations and liver biopsy.
Patient Management | 3 and 12 Months
  Confirmation at 3 months and at 12 months that recommended management at the index procedures was adequate.
Relationship between endoscopic findings on POCS visualization | 12 Months
  Relationship between endoscopic findings on POCS visualization during index procedure and refractory biliary strictures during follow-up.
Evaluation | 12 Months
  Evaluation by surgeon of whether or not POCS impacted patient management post procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Amrita Sethi, MD, Principal Investigator — Columbia University; Eduardo De Moura, MD, Principal Investigator — Hospital das Clinicas University of Sao Paulo; Adam Slivka, MD, Principal Investigator — University of Pittsburgh Medical Center; Andres Cardenas, MD, Principal Investigator — Hospital Clinic of Barcelona; Marco Bruno, MD, Principal Investigator — Erasmus Medical Center
Locations (5):
- United States (2):
  - New York Presbyterian Hospital CUMC, New York, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- Hospital das Clinicas, São Paulo, Brazil
- Erasmus Medical Center, Rotterdam, Netherlands
- Hospital Clinic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No